CLINICAL TRIAL: NCT02646982
Title: Candesartan's Effects on Alzheimer's Disease And Related Biomarkers
Acronym: CEDAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ihab Hajjar, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00084574; R01AG049752 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Results first posted 2022-09-29 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer's disease; hypertension medication; Mild Cognitive impairment; Amyloid Beta
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Plaque, Amyloid | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Candesartan (Experimental): Candesartan will be given orally once a day in a stepwise manner as follows: All participants will be initiated on 8 mg candesartan. The dose will be increased in 2 week increments to 16 mg and 32 mg as long as the systolic blood pressure (SBP) >100 mm Hg, diastolic blood pressure (DBP) >40 mm Hg and participant reports no symptoms of hypotension (dizziness or weakness). The highest achievable dose will be the Maximal Tolerated Dose (MTD) and the participant will receive this dose for the remaining duration of the study (participants will be treated for 1 year).
  Interventions: Drug: Candesartan
- Placebo (Placebo Comparator): Participants will receive a matched placebo once a day orally for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — A matched placebo will be given once daily for 12 months.
  Arms: Placebo
Drug: Candesartan — Candesartan will be started at 8 mg orally, once daily. The dose will be increased in 2 week increments to 16 mg and 32 mg orally, once a day, as long as SBP>100 mm Hg, DBP>40 mm Hg and there are no reported symptoms of hypotension (dizziness or weakness). Candesartan will be given for a total of 12 months.
  Other Names: Atacand
  Arms: Candesartan

SUMMARY:
This study is intended to investigate the safety of candesartan, a blood pressure medication, in non-hypertensive individuals who have mild cognitive impairment (MCI) due to Alzheimer's disease and its effect on disease biomarkers.

DETAILED DESCRIPTION:
This is a double-blind placebo-control randomized clinical trial that compares candesartan to placebo in individuals with mild cognitive impairment (MCI) who also have positive Alzheimer's Disease (AD) biomarkers. The investigators will assess if blocking the effect of Ang II using angiotensin receptor blockers (ARBs) is safe in non hypertensive MCI individuals and whether the use of candesartan will be associated with changes in cerebrospinal fluid disease biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment, defined by:

  * Subjective memory concern
  * Abnormal memory function documented using the Logical Memory subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale-Revised (the maximum score is 25): [<11 for 16 or more years of education; <9 for 8-15 years of education; <6 for <7 years of education]
  * Montreal Cognitive Assessment (MoCA) < 26
  * Clinical Dementia Rating scale /Memory sum Box score=0.5
  * General functional performance sufficiently preserved (Functional Assessment Questionnaire<9)
* Amyloid positivity determined by measuring the amyloid content in the brain. This can be determined by either cerebrospinal fluid (CSF) amyloid level or an amyloid scan (PIB-PET)

Exclusion Criteria:

* Intolerance to ARBs
* Current use of ARBs, angiotensin-converting enzyme inhibitors (ACEIs) (use of antihypertensive medications other than ACEI or ARBs for other indications is allowed)
* Current diagnosis of hypertension or current use of antihypertensive medication that is prescribed specifically for hypertensive therapy
* SBP less than 110 or DBP less than 40 mm Hg
* Renal disease (Creatinine >2.0 mg/dl), hyperkalemia (K>5.5 meq/dl), platelets<50,000/μl, or international normalized ratio (INR)>1.9
* Active medical or psychiatric diseases that in the judgment of the investigator would affect the safety of the subject or scientific integrity of the study
* Uncontrolled congestive heart failure reflected by poor exercise tolerance and shortness of breath
* History of stroke in the past 3 years
* Inability to have MRI (eg metal implants or cardiac pacemaker) with an exception for those who cannot have an MRI, if all other parts of the study are obtained successfully they may still be enrolled in the study, or cognitive assessment or inability to assess amyloid positivity (no lumbar puncture and no amyloid scan)
* History of increased intracranial pressure (ICP) or bleeding diathesis (from disease states or from use of anticoagulants such as warfarin, heparin and related products, rivaroxaban or Xarelto, apixaban or Eliquis, edoxaban or Savaysa, dabigatran or Pradaxa)
* Women of childbearing potential (non-menopausal)
* In those who are unable to demonstrate that they understood the details of the study (ie lack of decisional-capacity to consent), a study partner/surrogate who can sign on their behalf will be required, otherwise they will be excluded
* Current use of Lithium, as candesartan may increase lithium concentration to toxic levels

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-06-30; Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Hajjar, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Wesley Woods Center, Atlanta, Georgia

REFERENCES:
- [Derived] Hajjar I, Okafor M, Wan L, Yang Z, Nye JA, Bohsali A, Shaw LM, Levey AI, Lah JJ, Calhoun VD, Moore RH, Goldstein FC. Safety and biomarker effects of candesartan in non-hypertensive adults with prodromal Alzheimer's disease. Brain Commun. 2022 Oct 25;4(6):fcac270. doi: 10.1093/braincomms/fcac270. eCollection 2022. PMID 36440097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Wesley Woods Health Center of Emory Healthcare in Atlanta, Georgia, USA. Participant enrollment began June 30, 2016 and all follow up was complete by August 17, 2020.
Groups:
- Candesartan: Participants receiving candesartan given orally once a day in a stepwise manner. Participants were initiated on 8 mg candesartan. The dose was increased in 2 week increments to 16 mg and 32 mg, as tolerated. The highest achievable dose was the Maximal Tolerated Dose (MTD) and the participant received this dose for the remaining duration of the study (12 months total).
- Placebo: Participants receiving a placebo to match candesartan once a day orally for 12 months.
Period: Overall Study
Arm/Group | Candesartan | Placebo
Started | 38 | 39
Completed | 35 | 37
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Candesartan | Placebo | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.4) | 69.5 (8.5) | 68.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 36 | 39 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 30 | 32 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 39 | 77
Sitting Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 124.7 (13.6) | 126.7 (13.2) | 125.4 (13.5)
Sitting Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 67.9 (9.9) | 69.8 (10.1) | 68.8 (10.4)
Sitting Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 66.3 (11.1) | 67.3 (11.5) | 66.8 (11.2)
Montreal Cognitive Assessment (MoCA) Score [Mean (Standard Deviation); unit: score on a scale] — MoCA is an instrument to screen for mild cognitive dysfunction, assessing the cognitive domains of attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Total scores range from 0 to 30 with higher scores indicating better cognitive function. A normal score is considered to be 26 or higher.
  score on a scale | 20.9 (3.9) | 20.7 (2.7) | 20.8 (3.3)
Number of Participants Taking Cholinesterase inhibitors or Memantine [Count of Participants; unit: Participants] | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Hypotensive Episode
Description: Hypotension is defined as blood pressure <100/40 mm Hg. Blood pressure was measured according to the American Heart Association guidelines with the subject in the sitting position and rested for 5 minutes. An appropriate cuff size (covering 60% of upper arm length and 80% of arm circumference) was used and correct cuff placement (1-2 inches above the brachial pulse on bare arm) was ensured.
Time Frame: Up to Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
Participants | 16 | 4

2. Primary Outcome: Number of Participants With Symptoms of Hypotension
Description: Participants were asked to report any symptoms of hypotension (dizziness, weakness, fatigue and lightheadedness). All participants were given a telephone number to reach physician 24-hours per day to report symptoms they experience. The number of participants reporting symptoms of hypotension is reported here.
Time Frame: Up to Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
Participants | 7 | 10

3. Primary Outcome: Number of Participants With Hypotensive Episodes and Symptoms
Description: The number of participants with reported episodes hypotension as well as symptoms of hypotension.
Time Frame: Up to Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
Participants | 4 | 1

4. Primary Outcome: Number of Participants With Elevated Serum Creatinine
Description: The levels of creatinine were obtained from blood samples. Elevated serum creatinine is defined as levels >2.5 milligram per deciliter (mg/dL). Elevated serum creatinine is indicative of decreased renal function.
Time Frame: Up to Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Hyperkalemia
Description: The levels of potassium were obtained from blood samples. Hyperkalemia is defined as potassium levels >5.9 milliequivalent per deciliter (meq/dL). Hyperkalemia is an indication of kidney dysfunction.
Time Frame: Up to Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
Participants | 0 | 1

6. Primary Outcome: Number of Participants Discontinuing Study Medication
Description: The number of participants who discontinued the study medication is presented here.
Time Frame: Up to Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
Participants | 0 | 1

7. Secondary Outcome: Cerebrospinal Fluid (CSF) Total Tau Levels
Description: CSF total tau (t-tau) levels were analyzed from CSF samples obtained via lumbar puncture. Normal values for t-tau are < 450 pg/ml. Elevated levels of t-tau indicate worsening disease.
Time Frame: Baseline, Month 12
Population: This analysis includes participants who had CSF samples collected.
Measure: Least Squares Mean (Standard Error); unit: Picograms per milliliter (pg/ml)
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 36 | 37
Picograms per milliliter (pg/ml)
  Baseline Total Tau | 638.31 (53.61) | 529.04 (53.50)
  Month 12 Total Tau | 571.96 (52.89) | 441.25 (53.02)

8. Secondary Outcome: Cerebrospinal Fluid (CSF) of Tau Phosphorylated at Threonine 181 (p-tau181) Levels
Description: CSF levels of p-tau181 were analyzed from CSF samples obtained via lumbar puncture. P-tau181 is a biomarker that is elevated in persons with Alzheimer's disease. Higher values indicate worsening disease.
Time Frame: Baseline, Month 12
Population: This analysis includes participants who had CSF samples collected.
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 36 | 37
pg/ml
  Baseline p-tau | 100.29 (9.09) | 81.58 (9.07)
  Month 12 p-tau | 88.52 (8.58) | 68.49 (8.59)

9. Secondary Outcome: Cerebrospinal Fluid (CSF) Amyloid Aβ42 Levels
Description: CSF Aβ42 levels were analyzed from CSF samples obtained via lumbar puncture. Aβ42 is a biomarker for Alzheimer's disease and lower values indicate worsening disease and an increased accumulation of amyloid in the brain.
Time Frame: Baseline, Month 12
Population: This analysis includes participants who had CSF samples collected.
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 36 | 37
pg/ml
  Baseline Aβ42 | 554.80 (34.09) | 523.03 (33.98)
  Month 12 Aβ42 | 557.60 (27.32) | 476.32 (27.43)

10. Secondary Outcome: Cerebrospinal Fluid (CSF) Amyloid Aβ40 Levels
Description: CSF Aβ40 levels were analyzed from CSF samples obtained via lumbar puncture. Lower values indicate worsening disease and an increased brain accumulation of amyloid.
Time Frame: Baseline, Month 12
Population: This analysis includes participants who had CSF samples collected.
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 36 | 37
pg/ml
  Baseline Aβ40 | 11624.00 (625.86) | 10802.00 (623.82)
  Month 12 Aβ40 | 11769.00 (571.54) | 9735.00 (573.74)

11. Secondary Outcome: Cerebrospinal Fluid (CSF) Amyloid Aβ42/Aβ40 Levels
Description: CSF Aβ42/Aβ40 levels were analyzed from CSF samples obtained via lumbar puncture. A lower ratio indicates worsening disease.
Time Frame: Baseline, Month 12
Population: This analysis includes participants who had CSF samples collected.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 36 | 37
Ratio
  Baseline Aβ42/Aβ40 ratio | 0.049 (0.003) | 0.052 (0.003)
  Month 12 Aβ42/Aβ40 ratio | 0.050 (0.003) | 0.051 (0.003)

12. Secondary Outcome: Pulse Wave Velocity (PWV)
Description: Arterial stiffness was assessed by Pulse Wave Velocity (PWV). PWV is calculated as PWV=distance (d)/time (t) and the unit of measure is reported as meters per second (m/s). Lower values indicate a preferable measurement of arterial stiffness.
Time Frame: Baseline, Month 12
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
m/s
  Baseline | 7.81 [7.12 to 8.51] | 8.73 [8.05 to 9.40]
  Month 12 | 7.71 [7.03 to 8.40] | 8.14 [7.47 to 8.81]

13. Secondary Outcome: Augmentation Index (AI)
Description: Arterial stiffness was assessed by Augmentation Index (AI). The AI is a ratio measure of augmentation of central arterial pressure reflected in a pulse wave; the value is multiplied by 100 to provide a percentage. AI increases with age and is higher in persons with cardiovascular disease states. A lower value indicates a preferable state of arterial stiffness.
Time Frame: Baseline, Month 12
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of arterial stiffness
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
percentage of arterial stiffness
  Baseline | 29.95 [25.92 to 33.98] | 31.22 [27.24 to 35.20]
  Month 12 | 28.36 [24.45 to 32.27] | 26.66 [22.81 to 30.51]

14. Secondary Outcome: Hippocampal Volume
Description: Structural MRI images were acquired in order to assess hippocampal volume. Decreased hippocampal volume suggests neurodegenerative changes
Time Frame: Baseline, Month 12
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
mm^3
  Baseline | 6949.82 (151.66) | 6662.21 (151.49)
  Month 12 | 6761.12 (151.42) | 6521.30 (152.14)

15. Secondary Outcome: Vasoreactivity
Description: Cerebrovascular reactivity (CVR) is assessed with blood oxygenation level-dependent (BOLD) MRI. Vasoreactivity (VR) is the degree of change in BOLD signal relative to change in end tidal CO2. CVR is an indicator of microvascular function (higher indicates better function)
Time Frame: Month 12
Measure: Least Squares Mean (95% Confidence Interval); unit: (ml/100g/min)/mmHg
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
(ml/100g/min)/mmHg | 0.27 [0.006 to 0.53] | -0.17 [-0.42 to 0.08]

16. Secondary Outcome: Global Standardized Uptake Value Ratio (SUVR) of (11)C-Pittsburgh Compound B ((11)C-PiB)
Description: In-vivo amyloid imaging with positron emission tomography (PET) was conducted after intravenous administration of 15±1.5 millicurie (mCi) of the radiotracer (11)C-PiB. SUVR is a ratio of PET uptake measured in the brain region of interest and a disease free reference region. A higher SUVR is an indication of increased PET radiotracer uptake and worsening disease.
Time Frame: Baseline, 12 Months
Measure: Mean (95% Confidence Interval); unit: Ratio of target and reference regions
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
Ratio of target and reference regions
  Baseline | 1.32 [1.23 to 1.40] | 1.42 [1.32 to 1.52]
  Month 12 | 1.34 [1.23 to 1.45] | 1.46 [1.34 to 1.59]

17. Secondary Outcome: Global Standardized Uptake Value Ratio (SUVR) of [18F]T807
Description: In-vivo tau-PET imaging was conducted using the radiotracer [18F]T807. SUVR is a ratio of PET uptake measured in the brain region of interest and a disease free reference region. A higher SUVR is an indication of increased PET radiotracer uptake and worsening disease.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Error); unit: Ratio of target and reference regions
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
Ratio of target and reference regions
  Baseline | 1.33 (0.05) | 1.36 (0.04)
  Month 12 | 1.34 (0.06) | 1.34 (0.05)

18. Secondary Outcome: Clinical Dementia Rating (CDR) Score
Description: The CDR rates each of the six general domains involving memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care. An overall score, ranging from 0 to 3, can be calculated. A score of 0 = normal, 0.5 = very mild dementia, 1 = mild dementia, 2 = moderate dementia, and 3 = severe dementia.
Time Frame: Baseline, Month 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
score on a scale
  Baseline | 1.86 (0.15) | 1.85 (0.14)
  Month 12 | 2.18 (0.28) | 2.21 (0.27)

19. Secondary Outcome: EXecutive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER) Toolbox Composite Score
Description: The EXAMINER toolbox battery includes 11 tasks that generate 15 primary variables. Within this set, the EXAMINER includes working memory, inhibition, set shifting, and fluency. The parts of EXAMINER that were used for this study include: Flanker task (inhibition) which involves responding to a central stimulus while ignoring flanking stimuli that are either compatible or incompatible with the central stimulus; Set-shifting, a measure of mental flexibility; Spatial 1-Back test assesses spatial working memory; Dot Counting test assesses verbal working memory; Verbal Fluency tested using a List Generation test which require the participant to generate words beginning with a specific letter, and category fluency in which the participant generates words from a specified category (e.g., animals, fruits). A composite score is calculated where scores range from -1 to +1 and higher are reflective of better executive function.
Time Frame: Baseline, Month 6, Month 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
score on a scale
  Baseline | 0.03 (0.11) | -0.05 (0.11)
  Month 6 | 0.18 (0.14) | 0.04 (0.14)
  Month 12 | 0.07 (0.14) | -0.06 (0.14)

20. Secondary Outcome: Hopkins Verbal Learning Test (HVLT) Delayed Recall Score
Description: The Hopkins Verbal Learning Test (HVLT) is used to assess memory domains. Participants are read a list of 12 words and are asked to recall as many as they can remember. This is repeated for 3 trials followed by a 20 minute delay, and then participants are asked to recall as many words as they can. The delayed recall score ranges from 0 to 12 and higher scores indicate better memory.
Time Frame: Baseline, Month 6, Month 12
Measure: Least Squares Mean (Standard Error); unit: number of words recalled
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
number of words recalled
  Baseline | 4.83 (0.53) | 5.29 (0.52)
  Month 6 | 5.40 (0.52) | 5.08 (0.51)
  Month 12 | 5.10 (0.52) | 5.39 (0.51)

21. Secondary Outcome: Trail Making Test (TMT) Part B
Description: The Trail Making Test assesses executive function. In Part B of the TMT participants connect circles labeled with letters and numbers, in ascending order. The score is the amount of time it takes for the participant to complete the task. The average time is 75 seconds and times greater than 273 seconds indicate a deficit with executive function.
Time Frame: Baseline, Month 6, Month 12
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
seconds
  Baseline | 149.44 (14.00) | 142.93 (13.88)
  Month 6 | 122.04 (13.49) | 152.91 (13.35)
  Month 12 | 148.06 (16.01) | 152.96 (15.65)

22. Secondary Outcome: Trail Making Test (TMT) Part B - A
Description: In Parts A and B of the TMT, participants connect circles labeled with numbers, in ascending order. The score is the amount of time (in seconds) it takes for the participant to complete the task. The TMT Part A score reflects visuoperceptual abilities, and subtracting the score for Part A from the score from Part B (Part B-A, in seconds) provides a more accurate assessment of executive function. A lower score indicates greater executive function.
Time Frame: Baseline, Month 6, Month 12
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 38 | 39
seconds
  Baseline | 108.08 (14.06) | 91.56 (13.87)
  Month 6 | 81.59 (11.56) | 102.38 (11.45)
  Month 12 | 103.64 (13.90) | 103.50 (13.52)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected for the duration of each participant's study enrollment, from the time that individuals gave consent to participate through their final study visit (up to 12 months).
Arm/Group | Candesartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 20/38 | 17/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan (N=38) | Placebo (N=39)
Dizziness (General disorders) | 6 | 5
Fatigue, tiredness, weakness (General disorders) | 4 | 4
Headache (General disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Lightheadedness (General disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Pain at back of head (General disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Vasovagal syncope (General disorders) | 1 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Runny nose (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT02646982/Prot_SAP_002.pdf
  • Informed Consent Form (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT02646982/ICF_001.pdf